CLINICAL TRIAL: NCT04545086
Title: Effectiveness of Video Based Education Versus Music Therapy on Anxiety, Experience, and Co-operation Among Patients Undergoing Magnetic Resonance Imaging in Radiology Department at ILBS, New Delhi.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3/19
Record Dates: First submitted 2020-08-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-01

CONDITIONS: Effectiveness of Video Based Education Versus Music Therapy on Anxiety, Experience, and Co-operation Among Patients Undergoing Magnetic Resonance Imaging
Keywords: Anxiety, Video Based Education, Music Therapy, Experience, Cooperation, Magnetic Resonance Imaging
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants were assigned randomly to three groups
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VBE Group (Experimental): Video Based Education was given before undergoing MRI procedure and Anxiety was assessed within 20 minutes of Intervention. Assessment of Experience, Co-operation and Opinion regarding intervention was done.
  Interventions: Behavioral: Video Based Education, Music Therapy
- MT Group (Experimental): Music Therapy was given before undergoing MRI procedure and Anxiety was assessed within 20 minutes of Intervention. Assessment of Experience, Co-operation and Opinion regarding intervention was done.
  Interventions: Behavioral: Video Based Education, Music Therapy
- Control Group (No Intervention): Routine Information was given before undergoing MRI procedure and Anxiety was assessed within 20 minutes of Intervention. Assessment of Experience, Co-operation was done.

INTERVENTIONS:
Behavioral: Video Based Education, Music Therapy — Video Based Education and Music Therapy was given as a part of Interventions to relieve anxiety of patients undergoing Magnetic Resonance Imaging
  Other Names: VBE, MT
  Arms: MT Group; VBE Group

SUMMARY:
A study to assess the Effectiveness of Video Based Education Versus Music Therapy on Anxiety, Experience, and Co-operation among Patients undergoing Magnetic Resonance Imaging. This is a Experimental Multiple Interventions Pre test - Post test Design. Three groups namely, Video Based Education group, Music Therapy Group and control groups are there in study.There will be significant difference in the Mean Anxiety Scores, Experience level, and Co-operation level of patients undergoing MRI in Video Based Education , Music Therapy group and Control Group

ELIGIBILITY:
Inclusion Criteria:

* undergoing MRI with or without contrast
* having age between 18- 60 years.
* alert, oriented
* able to comprehend, speak and listen English or Hindi.
* patients without hearing and visual impairment.
* available during period of data collection

Exclusion Criteria:

* unconscious
* critically ill and sedated.
* visiting Radiology Department for other procedures such as Computed Tomography scan, and MRI brain
* having pain score of 3-10 on universal pain assessment scale..

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
to assess the effectiveness of Video Based Education Versus Music Therapy on Anxiety, Experience, and Cooperation among patients undergoing Magnetic Resonance Imaging | 45 minutes to 1 hour.
  State Trait Anxiety Inventory-state form (STAI-S) scale, Patients' Scan Experience Scale and Cooperation Scale for MRI Procedure respectively will be use

CONTACTS AND LOCATIONS:
Locations (1):
- Deepika Bist, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided